CLINICAL TRIAL: NCT02184689
Title: Efficacy and Safety of Fexinidazole in Children at Least 6 Years Old and Weighing Over 20 kg With Human African Trypanosomiasis (HAT) Due to T.b. Gambiense: a Prospective, Multicentre, Open Study, plug-in to the Pivotal Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNDiHATFEX006
Record Dates: First submitted 2014-06-19; First posted 2014-07-09 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Human African Trypanosomiasis (HAT)
MeSH Terms: interventions — fexinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fexinidazole (Experimental)
  Interventions: Drug: fexinidazole

INTERVENTIONS:
Drug: fexinidazole

SUMMARY:
The aim of the study is to assess the efficacy and safety of an oral regimen of fexinidazole (once daily for 10 days) in the treatment of stage 1 and stage 2 T.b. gambiense sleeping sickness in children at least 6 years old and over 20 kg bodyweight.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed by one of the parents or the child's legal representative
* Child assent to participate in the study collected in the presence of an impartial witness
* Age between 6 and 15 years old
* > 20 Kg bodyweight
* Boy or girl
* Able to ingest at least one complete meal per day (or at least one Plumpy'Nut® sachet)
* Able to swallow 600mg fexinidazole tablets
* Karnofsky index > 50
* Presence of trypanosomes in blood and/or lymph and/or CSF
* Permanent address and ability to comply with follow-up visit schedule

Exclusion Criteria:

* Child refusing to be included in the trial
* Bodyweight < 20 Kg
* Severe malnutrition, defined as having a BMI below 16 (- 2 Z-score of the norm according to WHO 2007 Growth reference data)
* Inability to take oral medication
* Pregnancy or breastfeeding
* Clinically relevant medical condition other than HAT that, in the Investigator's opinion, may jeopardize subject safety or interfere with participation in the study, including but not limited to significant liver or cardiovascular disease, active documented or suspected infection, central nervous system (CNS) trauma or seizure disorders, coma or altered consciousness
* Severely deteriorated general condition, such as cardiovascular shock, respiratory distress, or terminal illness
* Any medical condition (except HAT-specific symptoms) hindering communication with the Investigator as required for the completion of this study
* Any contraindication to imidazole products (known hypersensitivity to imidazoles)
* History of HAT treatment in the past 2 years
* Patients previously enrolled in the study or having already received fexinidazole.
* Expected follow-up difficulties (migrants, refugees, itinerant vendors, etc.).
* Current alcohol or drug abuse
* Clinically significant abnormal laboratory findings, including ASAT and/or ALAT > 2 times ULN // Total bilirubin > 1.5 times ULN // Severe leukopenia (< 2000/mm3) // Potassium (K+) < 3.5 mmol // Any other clinically significant abnormal laboratory value (see details in Investigator Manual)
* Pregnancy confirmed by a positive urine pregnancy test obtained within 24 hours (h) prior to start of study treatment (see Section 5.8.3 Contraception; p36) for girls over 12 years old and over
* ECG abnormalities assessed by a central cardiologist
* QTcF≥ 450 ms, as measured automatically (if first measurement is abnormal, a second assessment will be done at least 10-20 min later, with the patient in resting position).
* Patients not tested for malaria and/or not treated adequately for this infection
* Patients not treated adequately for soil transmitted helminthic diseases

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2014-05-03 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Outcome (success or failure) at the test of cure (ToC) | 12 months after the end of treatment
  Success at 12 months, adapted from the WHO criteria (51), is defined as a cured patient:
  * Patient alive;
  * AND no evidence of trypanosomes in any body fluid;
  * AND WBC ≤20/µL in CSF.

CONTACTS AND LOCATIONS:
Locations (1):
- Kinshasa, Democratic Republic of the Congo

REFERENCES:
- [Derived] Kande Betu Kumesu V, Mutombo Kalonji W, Bardonneau C, Valverde Mordt O, Ngolo Tete D, Blesson S, Simon F, Delhomme S, Bernhard S, Nganzobo Ngima P, Mahenzi Mbembo H, Fina Lubaki JP, Lumeya Vuvu S, Kuziena Mindele W, Ilunga Wa Kyhi M, Mandula Mokenge G, Kaninda Badibabi L, Kasongo Bonama A, Kavunga Lukula P, Lumbala C, Scherrer B, Strub-Wourgaft N, Tarral A. Safety and efficacy of oral fexinidazole in children with gambiense human African trypanosomiasis: a multicentre, single-arm, open-label, phase 2-3 trial. Lancet Glob Health. 2022 Nov;10(11):e1665-e1674. doi: 10.1016/S2214-109X(22)00338-2. Epub 2022 Sep 27. PMID 36179736